CLINICAL TRIAL: NCT02538770
Title: The Impact of Respiratory Pathogen PCR Assay on Treatment of Adult Patients: A Randomized Controlled Trial
Brief Title: Rapid Viral Diagnostics in Adults to Reduce Antimicrobial Consumption and Duration of Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PPSHP93/2014
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Respiratory Virus Infection; Fever of Unknown Origin; Dyspnea; Chest Pain
MeSH Terms: conditions — Fever of Unknown Origin; Dyspnea; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid Anyplex TMII RV16 Detection (Experimental): Intervention is the rapid performance of Anyplex TMII RV16 detection
  Interventions: Other: Rapid diagnostics using Anyplex TMII RV16 Detection
- Delayed Anyplex TMII RV16 Detection (Active Comparator): Comprative intervention is the delayed performance of Anyplex TMII RV16 detection
  Interventions: Other: Delayed diagnostics Anyplex TMII RV16 Detection

INTERVENTIONS:
Other: Rapid diagnostics using Anyplex TMII RV16 Detection — Rapid diagnostics using Anyplex TMII RV16 Detection, i.e. physician receives results of respiratory virus PCR as soon as they are available
  Arms: Rapid Anyplex TMII RV16 Detection
Other: Delayed diagnostics Anyplex TMII RV16 Detection — Delayed diagnostics Anyplex TMII RV16 Detection, i.e. physician receives results of respiratory virus PCR after one week delay unless specifically solicited
  Arms: Delayed Anyplex TMII RV16 Detection

SUMMARY:
Viral respiratory infections are common and often require use of health care resources. Patients receive inappropriate bacterial antibiotics, which has many problems including side-effects, development of resistance and costs.

A small portion of the infections leads to severe clinical manifestations including hospitalisations and deaths. The significance of influenza virus is well known and it is actively detected in all age groups. However, the benefits of detecting other respiratory viruses have mainly been studied among children but not among adults. The development of multiplex PCR technique has provided a new and sensitive method for diagnosing a large panel of viruses. To convince the economical benefits of the rapid viral diagnostic in adult infectious patient, more evidence is needed.

In our randomized study, nasal and pharyngeal samples from the patients evaluated at the emergency clinic of internal medicine in the University Hospital of Oulu because of any respiratory symptom, chest pain or fever, will be collected. The samples will be tested for 16 different respiratory viruses by using Anyplex TMII RV16 Detection. The adult participants will be randomized in two groups. In one group the results of the testing will be reported for the attending physician as soon as possible, and in the other group 7 days after sampling. The effect of this delay to patient care is monitored. Also the results of children and adults are compared as well as results of men and women. The hypothesis is that rapid viral diagnostics shortens the length of admission and diminishes the use of bacterial antibiotics. New information on the viral epidemiology among children and adults is provided and clinical manifestations of specific viral infections in adults are described.

The estimated 1500 samples are also tested for 5 different respiratory bacteria by Anyplex TM II RB5 Detection. These results will be examined after completion of the study period. The benefits of rapid bacterial detection are evaluated in respect to the clinical course of the disease and considering the infection control aspects as well.

DETAILED DESCRIPTION:
Aim and Hypothesis

The aim of the study is:

1. To find out how the modern rapid multiplex-PCR based respiratory virus detection method affects the patient care
2. To examine does it shorten the length of admission and reduce antibiotic consumption
3. Compare the seasonality of different viruses in children and adults
4. Investigate the development and progress of an epidemic
5. Study the differences in the prevalence and severity of infections between genders
6. Describe clinical manifestations of different viral infections in adults
7. View more closely certain subgroups such as patients with chest pain in respect to different viral epidemics and their effect on the hospital admission rates
8. Evaluate the information provided by the bacterial detection

Subjects Our hospital is both a regional and a university hospital at the same time. Patients come to our clinic from a quite large area surrounding the city of Oulu and they represent the general population of the area well. The study population will be recruited 2014-2015 in the emergency clinics for pediatric and internal medicine patients in the Oulu University Hospital. Participants are patients with respiratory infection symptoms, chest pain or fever. Fever is determined as body temperature of 38 degrees centigrade or more measured either in the hospital or at home.

Study design This is a randomized clinical trial evaluating the impact of modern multiplex PCR based respiratory virus diagnostics on treatment and outcome of adult patients. Participants are randomized in two groups with results being reported either immediately or after a week (Picture 1). In children the viral PCR diagnostics is already routinely used and collection of nasal and pharyngeal samples continues normally. All pediatric results are reported immediately. Approval of the ethical review board of the Northern Ostrobothnia Hospital District has been acquired.

Course of the study Data collection All patients entering the internal medicine emergency clinics because of respiratory infection symptoms (cough, rhinitis, shortness of breath, sore throat), chest pain or fever will be given the opportunity to participate in the study. After signing an informed consent a nasal and a pharyngeal swab will be taken for viral examination. Adult patients are randomized in two different groups. In one group the results of the viral detection are reported immediately and in the other group they are reported 7 days after sampling.

Samples will be analyzed in the microbiological laboratory by real time PCR method Anyplex TMII to detect genome of 16 different respiratory viruses and of 5 different bacterial pathogen (Table 1). Results in the delayed group will be given earlier in the case the clinician is requesting them. The results of the bacterial findings will be analyzed after completion of the study since the clinical relevance of them is not clear yet. The bacteriological diagnostic of the patients during the study relies on the routinely used methods.

The attending clinician decides the treatment and care of the patient independently. Patient's chart will be reviewed for the course of disease, antibiotic use, ICU care and length of hospital stay. The results of key laboratory tests and microbiological findings will be collected. Radiological findings will be registered. At discharge, the participants are asked to report the duration of the symptoms, absence from work and the date of a possible doctors follow up. The population register centre will be used at the end of the study to find out the number of deceased, and their time and cause of the death will be recorded

. Table 1. Microbes detected from the study samples Viruses (AnyplexTMII RV16 Detection) Adenovirus Influenza A/B virus Parainfluenza virus1/2/3/4 Rhinovirus A/B/C Respiratory syncytial virus A/B Bocavirus 1/2/3/4 Metapneumovirus Coronavirus 229E/NL63/OC43 Enterovirus

Data analysis The length of hospital admission and the use of bacterial antibiotics is compared between the randomized groups. Viral findings of children and adults will be evaluated. The emergence of viruses in different areas of the district as well as in different age groups is examined. The differences in clinical picture and in microbiological findings between genders are viewed. The symptoms and clinical findings in adults with detected RSV or metapneumovirus are described. The bacterial findings are evaluated and compared with clinical data to determine the significance of the information provided by the test.

Impact of the study In our hospital major part of the viral respiratory infection diagnostics in adults has been accomplished by influenza virus antigen detection. Now a more sensitive measure for detecting 16 different respiratory pathogens from nasopharyngeal sample is available. We will determine whether more specific identification of the etiological agent affects the patient care. If the accurate diagnostics diminishes inappropriate antibiotic use it saves the patient from potential side effects and the society from unnecessary costs. Importantly it also saves the microbial flora from the antibiotic selection pressure which is considered to facilitate the emergence of antibiotic resistance. In children the benefits of accurate diagnostics have been recognized but in adults this is still under progress. This study is designed to demonstrate these advantages in adults.

ELIGIBILITY:
Inclusion Criteria:

* All patients visiting Oulu University Hospital emergency room or admitted to acute pulmonology ward AND signs of possible respiratory tract infection such as cough, fever or dyspnea OR chest pain

Exclusion Criteria:

* No exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization | One month
  The number of days in hospital within one month after randomization
Antimicrobial consumption | One month
  Number of days on antimicrobials within one month after randomization
Antimicrobial consumption | One month
  Defined daily doses of antimicrobial agents within one month after randomization

SECONDARY OUTCOMES:
Number of radiological examinations | One month
Cost of other examinations in hospital | One month

CONTACTS AND LOCATIONS:
Overall Officials: Marjo Renko, PhD, MD, Principal Investigator — Oulu University Hospital
Locations (2):
- Finland (2):
  - Emergency Room of Oulu University Hospital, Oulu
  - Pulmonology ward Oulu University Hospital, Oulu